CLINICAL TRIAL: NCT02312479
Title: Safety and Performance Study of the Use of the Nyxoah SAT System for the Treatment of Obstructive Sleep Apnea
Brief Title: Safety and Performance Study of the Nyxoah SAT System for Treating OSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nyxoah S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT2014A
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nyxoah SAT therapy (Experimental)
  Interventions: Device: Nyxoah SAT system

INTERVENTIONS:
Device: Nyxoah SAT system — The Nyxoah SAT system is comprised of an implantable nerve stimulator implanted over one of the tongue muscles via a minimally invasive procedure. Stimulation of the Hypoglossal nerves causes the tongue muscles to contract, thus maintaining an open airway during sleep.

SUMMARY:
A prospective open-label, single treatment study to assess the safety and the performance of the Nyxoah SAT system for the treatment of Obstructive Sleep Apnea

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate to severe Obstructive Sleep Apnea
* Have failed or have not tolerated CPAP treatment
* Willing and capable of providing informed consent
* Willing and capable of returning to all follow-up visits and sleep studies, including evaluation procedures and filling out questionnaires

Exclusion Criteria:

* BMI limits
* Subjects with complete concentric collapse at the soft palate level per endoscopy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence of serious device related adverse events | 6-months post-implantation
Mean change of AHI (Apnea-Hypopnea Index) measured by in-lab polysomnography (PSG) from baseline measurement to 6-months post-implantation | 6-months post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Joachim T Maurer, OA Dr. med., Principal Investigator — Universitäts-HNO-Klinik Mannheim; Evert Hamans, PhD Dr., Principal Investigator — Universiteit Antwerpen
Locations (2):
- Antwerp University Hospital, Edegem, Belgium
- Universitäts-HNO-Klinik Mannheim, Mannheim, Germany